CLINICAL TRIAL: NCT00374946
Title: A Randomised Controlled Clinical Study Ofbearing Surfaces in Four Hybrid Prosthesis - Results After 10 Years
Brief Title: A Clinical Evaluation of Wear Couples in THA
Status: Completed | Type: Observational
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Arne Borgwardt, MD Head of Department, Frederiksberg University Hospital
Other Study IDs: KF-01-355/98; NCT00289692 (obsolete NCT alias)
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Articular Bearing Surface Wear of Prosthetic Joint; Wear of Articular Bearing Surface of Prosthetic Joint; Prosthesis Survival
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: THA. Bearing of Zirconia head and UHMWPE liner
  Interventions: Device: THA
- B: THA. Bearing of CO-Cr-Mo head and liner
  Interventions: Device: THA
- C: THA. Head og Zirconia head and UHMWPE moulded in shell (Asian)
  Interventions: Device: THA
- D: THA. Head and shell og Alumina ceramic
  Interventions: Device: THA

INTERVENTIONS:
Device: THA

SUMMARY:
Clinical evaluation of 4 different bearings in THA. Primary parameter being prosthetic survival data.

ELIGIBILITY:
Inclusion Criteria:

* >18 Willing to participate informed consents indication for THA

Exclusion Criteria:

* <18 other diseases in the lower extremities than the actual disorder of the hip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the orthopedic department in the inclusion period fulfilling the inclusion criteria and not having any of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2000-12; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arne Borgwardt, md, Principal Investigator — Frederiksberg UH